CLINICAL TRIAL: NCT03877237
Title: International, Multicentre, Parallel-group, Randomised, Double-blind, Placebo-controlled, Phase III Study Evaluating the Effect of Dapagliflozin on Exercise Capacity in Heart Failure Patients With Reduced Ejection Fraction
Brief Title: DETERMINE-reduced - Dapagliflozin Effect on Exercise Capacity Using a 6-minute Walk Test in Patients With Heart Failure With Reduced Ejection Fraction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D169EC00002; 2018-003442-16 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-03-15 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF)
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Green, diamond shaped, film coated tablets 10 mg administered orally, once daily
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Green, diamond shaped, film coated tablets placebo administered orally, once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Tablets administered orally once daily. Treatment start within 24h after randomisation for 16 weeks.
  Arms: Dapagliflozin
Other: Placebo — Tablets administered orally once daily. Treatment start within 24h after randomisation for 16 weeks.
  Arms: Placebo

SUMMARY:
International, Multicentre, Parallel-group, Randomised, Double-blind, Placebo-controlled, Phase III Study Evaluating the effect of Dapagliflozin on Exercise Capacity in Heart Failure Patients with Reduced Ejection Fraction (HFrEF)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedures
* Male or female, aged ≥18 years
* Documented diagnosis of symptomatic HFrEF (NYHA functional class II-IV), which has been present for at least 8 weeks
* LVEF≤40%
* Elevated NT-proBNP levels
* Patients should receive background standard of care as described below: All HFrEF patients should be treated according to locally recognised guidelines on standard of care treatment with both drugs and devices, as appropriate. Guideline-recommended medications should be used at recommended doses unless contraindicated or not tolerated. Therapy should have been individually optimised and stable for ≥4 weeks (this does not apply to diuretics) before visit 1 and include (unless contraindicated or not tolerated):

  * an ACE inhibitor, or ARB or sacubitril/valsartan and
  * a beta-blocker and
  * if considered appropriate by the patient's treating physician; a mineral corticoid receptor antagonist
* 6MWD≥100 metres and ≤425 metres at enrolment and randomization.

Exclusion Criteria:

* Presence of any condition that precludes exercise testing
* Participation in a structured exercise training programme in the 1 month prior to screening or planned to start during the trial
* Receiving therapy with an SGLT2 inhibitor within 4 weeks prior to enrolment or previous intolerance of an SGLT2 inhibitor
* Type 1 diabetes mellitus
* eGFR <25 mL/min/1.73 m2 (CKD-EPI formula) at enrolment, unstable or rapidly progressing renal disease at time of randomisation
* Systolic BP <95 mmHg on 2 consecutive measurements
* Systolic BP ≥160 mmHg if not on treatment with ≥3 blood pressure lowering medications or ≥180 mmHg irrespective of treatments, on 2 consecutive measurements
* Current acute decompensated HF or hospitalisation due to decompensated HF <4 weeks prior to enrolment
* MI, unstable angina, coronary revascularization ablation of atrial flutter/fibrillation, valve repair/replacement, implantation of a cardiac resynchronization therapy device within 12 weeks prior to enrolment or planned to undergo any of these operations after randomization.
* Stroke or transient ischemic attack within 12 weeks prior to enrolment.
* Primary pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease including COPD.
* Previous cardiac transplantation or implantation of a ventricular assistance device or similar device, or implantation expected after randomization
* HF due to infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, cardiac tamponade, known genetic hypertrophic cardiomyopathy or obstructive hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy/dysplasia, or uncorrected primary valvular disease

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-03-07 (Actual); Study Completion 2020-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (69):
- United States (22):
  - Research Site, Alexander City, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Fort Payne, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Torrance, California
  - Research Site, Stamford, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Tucker, Georgia
  - Research Site, Munster, Indiana
  - Research Site, Petoskey, Michigan
  - Research Site, Kansas City, Missouri
  - Research Site, New Brunswick, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Rosedale, New York
  - Research Site, Burlington, North Carolina
  - Research Site, Abington, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Tullahoma, Tennessee
  - Research Site, Falls Church, Virginia
  - Research Site, Seattle, Washington
- Brazil (3):
  - Research Site, Blumenau
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (14):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Ajax, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Stoney Creek, Ontario
  - Research Site, York, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Georges, Quebec
- Denmark (10):
  - Research Site, Århus N
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Hellerup
  - Research Site, Hjørring
  - Research Site, Hvidovre
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Randers
  - Research Site, Svendborg
- Japan (8):
  - Research Site, Daito-shi
  - Research Site, Kobe
  - Research Site, Matsubara-shi
  - Research Site, Naha
  - Research Site, Osaka
  - Research Site, Sayama-shi,
  - Research Site, Shunan-shi
  - Research Site, Takarazuka-shi
- Slovakia (3):
  - Research Site, Lučenec
  - Research Site, Martin
  - Research Site, Prešov
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Diepkloof, Soweto
- South Korea (2):
  - Research Site, Gangwon-do
  - Research Site, Seoul
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Östersund
  - Research Site, Stockholm
  - Research Site, Umeå

REFERENCES:
- [Derived] Docherty KF, Buendia Lopez R, Folkvaljon F, de Boer RA, Cowie MR, Hammarstedt A, Kitzman DW, Kosiborod MN, Langkilde AM, Reicher B, Senni M, Shah SJ, Verma S, Solomon SD, McMurray JJV. Effect of Dapagliflozin on Accelerometer-Based Measures of Physical Activity in Patients With Heart Failure: An Analysis of the DETERMINE Trials. Circ Heart Fail. 2024 Oct;17(10):e012349. doi: 10.1161/CIRCHEARTFAILURE.124.012349. Epub 2024 Aug 30. PMID 39212948
- [Derived] McMurray JJV, Docherty KF, de Boer RA, Hammarstedt A, Kitzman DW, Kosiborod MN, Maria Langkilde A, Reicher B, Senni M, Shah SJ, Wilderang U, Verma S, Solomon SD. Effect of Dapagliflozin Versus Placebo on Symptoms and 6-Minute Walk Distance in Patients With Heart Failure: The DETERMINE Randomized Clinical Trials. Circulation. 2024 Mar 12;149(11):825-838. doi: 10.1161/CIRCULATIONAHA.123.065061. Epub 2023 Dec 7. PMID 38059368
- See also: redacted Clinical Study Protocol (CSP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169EC00002&attachmentIdentifier=d63ceb7a-2a2d-4a96-9adb-722a4237ce11&fileName=d169ec00002-csp-v2_Redacted.pdf&versionIdentifier=
- See also: redacted Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D169EC00002&attachmentIdentifier=7c255e2c-42d1-4f94-85b7-3724c96b4c0e&fileName=d169ec00002-sap-ed-3_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapa 10mg: Dapagliflozin 10 mg, given once daily per oral use.
- Placebo: Placebo tablet to match dapagliflozin 10 mg, given once daily per oral use.
Period: Overall Study
Arm/Group | Dapa 10mg | Placebo
Started | 156 | 157
Treated | 156 | 157
Completed | 151 | 151
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 2
Not completed — Death | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All participants that were randomized, regardless of whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapa 10mg | Placebo | Total
Number analyzed (Participants) | 156 | 157 | 313
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (9.84) | 67.3 (10.95) | 67.8 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 35 | 80
  Male | 111 | 122 | 233
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 21 | 39
  Not Hispanic or Latino | 138 | 136 | 274
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 100 | 98 | 198
  Black or African American | 25 | 22 | 47
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 27 | 46
  Other | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Kansas-City Cardiomyopathy Questionnaire-Total Symptom Score (KCCQ-TSS) at Week 16 (Higher Scores Represent Less HF Symptom Frequency and Burden).
Description: Change from baseline in KCCQ-TSS was defined as the endpoint value at week 16 minus the baseline value. KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ-TSS incorporates the symptom frequency (4 items) and symptom burden (3 items) domains into a single summary score. The score is transformed to a range of 0-100, in which a higher score reflects better health status. Baseline value is the last value on or prior to the randomization visit. Deaths are treated as the worst outcome and ordering among deaths is based on last value while alive. In rank ANCOVA and HL estimation, multiple imputation was performed on missing values for participants who were alive at the visit at week 16 but did not have KCCQ-TSS values.
Time Frame: At baseline and at week 16 or death before week 16
Population: Full Analysis Set: All participants that were randomized, regardless of whether treated or not.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Dapa 10mg | Placebo
Number analyzed (Participants) | 156 | 157
Score on a scale | 2.08 [-4.17 to 14.58] | 0.00 [-10.42 to 9.38]
Statistical Analysis 1: Comparison: Dapa 10mg vs Placebo; For the primary efficacy endpoint KCCQ-TSS, the following hypothesis was tested using the significance level 0.04990 * H0: m(r(A)) = m(r(C)) versus * H1: m(r(A)) ≠ m(r(C)) Where H0 and H1 are the null and alternative hypotheses, respectively, and m(r(A)) and m(r(C)) represent the median of the ranked changes in the primary efficacy endpoint, KCCQ-TSS, from baseline to week 16, among patients receiving dapagliflozin (Active) and placebo (Control) treatment, respectively; Test type: Superiority; p = 0.02164, Rank ANCOVA — To account for multiplicity, a pre-specified testing strategy was followed to control the overall type I error rate; Model includes baseline rank of outcome variable as a covariate, treatment group as a factor, and is stratified by T2DM status at randomization; Hodges-Lehmann median diff. vs placebo = 4.23, 95% CI 2-sided [0.96 to 8.22]

2. Primary Outcome: Change From Baseline in Kansas-City Cardiomyopathy Questionnaire-Physical Limitation Score (KCCQ-PLS) at Week 16 (Higher Scores Represent Less Physical Limitation Due to HF)
Description: Change from baseline in KCCQ-PLS was defined as the endpoint value at week 16 minus the baseline value. KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. The KCCQ-PLS incorporates the 6 physical limitation items into a single score. The score is transformed to a range of 0-100, in which a higher score reflects better health status. Baseline value is the last value on or prior to the randomization visit. Deaths are treated as the worst outcome and ordering among deaths is based on last value while alive. Deaths are treated as the worst outcome and ordering among deaths is based on last value while alive. In rank ANCOVA and HL estimation, multiple imputation was performed on missing values for participants who were alive at the visit at week 16 but did not have KCCQ-PLS values.
Time Frame: At baseline and at week 16 or death before week 16
Population: Full Analysis Set: All participants that were randomized, regardless of whether treated or not, excluding participants with non-calculable baseline or week 16 KCCQ-PLS.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Dapa 10mg | Placebo
Number analyzed (Participants) | 153 | 156
Score on a scale | 4.17 [-4.17 to 12.50] | 0.00 [-8.33 to 8.33]
Statistical Analysis 1: Comparison: Dapa 10mg vs Placebo; For the primary efficacy endpoint KCCQ-PLS, the following hypothesis was tested at significant level of 0.04990 * H0: m(r(A)) = m(r(C)) versus * H1: m(r(A)) ≠ m(r(C)) Where H0 and H1 are the null and alternative hypotheses, respectively, and m(r(A)) and m(r(C)) represent the median of the ranked changes in the primary efficacy endpoint, KCCQ-PLS, from baseline to week 16, among patients receiving dapagliflozin (Active) and placebo (Control) treatment, respectively; Test type: Superiority; p = 0.05842, Rank ANCOVA — KCCQ-PLS was tested at the alpha level of 0.04990 because KCCQ-TSS had a statistically significant p-value, in accordance with the pre-specified testing strategy; [statistical method as in outcome 1, analysis 1]; Hodges-Lehmann median diff. vs placebo = 4.17, 95% CI 2-sided [0.03 to 8.33]

3. Primary Outcome: Change From Baseline in 6-minute Walk Distance (6MWD) at Week 16 (Larger Distances Represent Better Functional Capacity).
Description: Change from baseline in 6-minute walk distance (6MWD) (exercise capacity) at week 16 was defined as the distance walked in 6 minutes at week 16 minus the baseline value. Baseline value is the last value on or prior to the randomization visit. Deaths are treated as the worst outcome and ordering among deaths is based on last value while alive. In rank ANCOVA and HL estimation, multiple imputation was performed on missing values for participants who were alive at the visit at week 16 but did not have 6MWD values.
Time Frame: At baseline and at week 16 or death prior to week 16
Population: Full Analysis Set: All participants that were randomized, regardless of whether treated or not.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Dapa 10mg | Placebo
Number analyzed (Participants) | 156 | 157
meters | 20.0 [-2.0 to 42.0] | 13.5 [-12.5 to 46.5]
Statistical Analysis 1: Comparison: Dapa 10mg vs Placebo; For the primary efficacy endpoint 6MWD, the following hypothesis was tested using the significance level 0.00010: H0: m(r(A)) = m(r(C)) versus H1: m(r(A)) ≠ m(r(C)) Where H0 and H1 are the null and alternative hypotheses, respectively, and m(r(A)) and m(r(C)) represent the median of the ranked changes in the primary efficacy endpoint, 6MWD, from baseline to week 16, among patients receiving dapagliflozin (Active) and placebo (Control) treatment, respectively; Test type: Superiority; p = 0.68626, Rank ANCOVA — To account for multiplicity, a pre-specified testing strategy was followed to control the overall type I error rate; [statistical method as in outcome 1, analysis 1]; Hodges-Lehmann median diff. vs placebo = 3.2, 95% CI 2-sided [-6.5 to 13.0]

4. Secondary Outcome: Change From Baseline at the End of the Study in the Total Time Spent in Light to Vigorous Physical Activity, as Assessed Using a Wearable Activity Monitor (Accelerometer).
Description: Change from baseline at the end of the study in total time spent in light to vigorous physical activity (LVPA), as assessed using a wearable activity monitor, was defined as the total time [per day] spent in LVPA at the end of the study minus the baseline value. Baseline is the 7 day period starting on the day of enrolment and ending before randomization. End of study is defined as the period starting on the day of week 14 and prior to the week 16 visit. Deaths are treated as the worst outcome and ordering among deaths is based on last value while alive.
Time Frame: At baseline and at end of study or death before week 16.
Population: Full Analysis Set: All participants that were randomized, regardless of whether treated or not, including participants from investigator sites having wearable activity monitor data collected.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dapa 10mg | Placebo
Number analyzed (Participants) | 42 | 34
hours | -0.19 [-0.57 to 0.15] | -0.15 [-0.68 to 0.53]
Statistical Analysis 1: Comparison: Dapa 10mg vs Placebo; For the secondary efficacy endpoint, total time spent in LVPA, the testing hypothesis is * H0: m(r(A)) = m(r(C)) versus * H1: m(r(A)) ≠ m(r(C)) Where H0 and H1 are the null and alternative hypotheses, respectively, and m(r(A)) and m(r(C)) represent the median of the ranked changes in secondary efficacy endpoint, total time spent in LVPA, from baseline to End of study among patients receiving dapagliflozin (Active) and placebo (Control) treatment, respectively; Test type: Superiority; p = 0.19748, Rank ANCOVA — Total time spent in LVPA was not tested for statistical significance and the p-value is considered nominal because the test for 6MWD was not statistically significant; [statistical method as in outcome 1, analysis 1]; Hodges-Lehmann median diff. vs placebo = -0.16, 95% CI 2-sided [-0.55 to 0.22]

ADVERSE EVENTS:
Time Frame: Includes data collected on or after date of first dose and up to (including) 30 days following last dose of randomized study drug, and no later than visit 5 (up to day 119). Deaths collected on or after first dose of randomized study drug, up to 119 days.
Description: For analysis of Adverse Events Safety analysis set is used. Safety analysis set : All randomized participants who received at least one dose of study drug.
Arm/Group | Dapa 10mg | Placebo
All-Cause Mortality (participants affected / at risk) | 3/156 | 2/157
Serious Adverse Events (participants affected / at risk) | 19/156 | 23/157
Other Adverse Events (participants affected / at risk) | 0/156 | 0/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dapa 10mg (N=156) | Placebo (N=157)
Cardiac failure (Cardiac disorders) | 3 | 6
Cardiac arrest (Cardiac disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 1 | 4
Left ventricular failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Chagas' cardiomyopathy (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Non-cadiac chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
In this study, a subset of participants received wearable activity monitors to wear at home for 3 periods of 7 days. Data collection from the wearable device was challenging and a substantial amount of data was missing. This limits the use of the data based on the wearable activity monitors to investigate the potential impact of study drug on the amount, duration, and intensity of physical activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03877237/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT03877237/SAP_001.pdf